CLINICAL TRIAL: NCT05342246
Title: Success Rates for Management of Separated Instruments in Canals With Type II Vertucci's Classification: Prospective Clinical Study
Brief Title: Success Rates for Management of Separated Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Mokhtar Nagy, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec IR012249
Record Dates: First submitted 2022-04-16; First posted 2022-04-22 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Teeth, Endodontically-Treated
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conservative treatment (Experimental): The patent canal is retreated, no attempt to deal with the separated instrument
  Interventions: Procedure: Endodontic retreatment
- traditional (Active Comparator): All canals are retreated with attempts to retrieve the broken file
  Interventions: Procedure: Endodontic retreatment

INTERVENTIONS:
Procedure: Endodontic retreatment — retreatment of the patent root canal only without attempt to retrieve the separated instrument

SUMMARY:
The study compares the prognosis of cases of Separated Instruments in Canals With Type II Vertucci's Classification treated with conservative approach

DETAILED DESCRIPTION:
Teeth with Type II Vertucci root canal configuration are having more incidence of instruments separation due the presence of an S-type (Double curve). The aim of this study is to compare the outcome of minimally invasive approach (MIA), retaining the separated in one root canal, cleaning and shaping of portals of entry of the two canals and portal of exit of both canals through the other patent canal, in comparison to the outcome of retrieval of the broken instrument by ultrasonics retrieval techniques (URT)

ELIGIBILITY:
Inclusion Criteria:

* Presence of separated instrument in a root with a Vertucci's type II configuration (the level of the SI was evaluated using CBCT scans)
* Age range 35-55 years
* Teeth having a baseline periapical lesion (PAI score ≥2) in the affected root

Exclusion Criteria:

* • Patients who refused to undergo radiographic follow-up.

  * Pregnant females.
  * Patients suffered from a systemic disease.
  * Teeth with lesions connected to adjacent teeth.
  * Teeth with root fractures or perforations.
  * Teeth with lesion communicating with the alveolar crest.
  * patients with generalized chronic periodontitis or teeth that need periodontal surgery prior to coronal restorations due to marginal deficiency
  * teeth with damaged or resorbed peri- apex
  * teeth that were treated with a fiber post and teeth with canal curvature more than 25 degrees

Ages: 33 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
monitoring of periapical index | 2 years
  The peri-radicular condition was evaluated using the Periapical Index (PAI) created by Ørstavik et al. (1986). The PAI includes five grades represented on an ordinal scale as follows: (1) normal periapical structures; (2) small changes in the periapical bone or bone structure; (3) changes in the periapical bone structure with mineral loss, characteristic of apical periodontitis; (4) demineralization of the periapical bone within a well-defined radiolucent area; and (5) demineralization of the periapical bone with exacerbations and expansion in bone structure.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hulsmann M. Methods for removing metal obstructions from the root canal. Endod Dent Traumatol. 1993 Dec;9(6):223-37. doi: 10.1111/j.1600-9657.1993.tb00278.x. PMID 8143573
- [Result] Ward JR, Parashos P, Messer HH. Evaluation of an ultrasonic technique to remove fractured rotary nickel-titanium endodontic instruments from root canals: an experimental study. J Endod. 2003 Nov;29(11):756-63. doi: 10.1097/00004770-200311000-00017. PMID 14651285